CLINICAL TRIAL: NCT06263114
Title: Correlation of Blood Gene Expression (TruGraf Liver) With Liver Biopsy in Pediatric Liver Transplant Recipients
Status: Terminated | Type: Observational
Why Stopped: Sponsor requested study closure
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Eurofins (Industry)
Responsible Party: Principal Investigator, Ryan Fischer, MD, Chief, Section of Hepatology and Transplant Medicine, Children's Mercy Hospital Kansas City
Other Study IDs: 00002826
Record Dates: First submitted 2024-02-07; First posted 2024-02-16 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Liver Transplant; Complications; Liver Failure, Acute
Keywords: Pediatric
MeSH Terms: conditions — Liver Failure, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: TruGraf® Liver gene expression panel (GEP) — Test done on blood sample collected during for cause or routine liver biopsy

SUMMARY:
Liver transplant rejection is when the body's immune system attacks and damages the liver of a transplant recipient. Currently the best way to see if that is happening is with a liver biopsy. The purpose of this research study is to see if a simple blood test can diagnose if a transplanted liver is being rejected.

DETAILED DESCRIPTION:
This study is an investigator-initiated, prospective, single-cohort trial to assess the ability of the TruGraf® Liver gene expression panel (GEP) to predict rejection in pediatric liver transplant recipients undergoing surveillance and for-cause liver biopsy.

ELIGIBILITY:
Inclusion Criteria:

• All liver transplant patients at least 1 year of age and less than 18 years of age undergoing surveillance or for-cause liver biopsy

Exclusion Criteria:

• Non-English, non-Spanish Speaking

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric Liver Transplant
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Correlation of the TruGraf® Liver GEP with rejection activity index (RAI) on surveillance and for-cause biopsy. | Week prior to or at time of biopsy
  To evaluate the performance of the blood-based TruGraf® Liver GEP to accurately diagnose rejection, confirmed by surveillance or for-cause liver biopsy.

SECONDARY OUTCOMES:
Comparison of the GEP to non-rejection injury found on biopsy | Week prior to or at time of biopsy
  A comparison of the GEP to non-rejection injury (e.g., infection) found on biopsy
Utility of the GEP for monitoring liver injury | Week prior to or at time of biopsy
  Utility of the GEP for monitoring liver injury (i.e., as treatment is weaned, does the GEP return to a non-rejection correlate).

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Fischer, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospitals and Clinics, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be available

DOCUMENTS (2):
  • Study Protocol (2023-01-03): https://cdn.clinicaltrials.gov/large-docs/14/NCT06263114/Prot_000.pdf
  • Informed Consent Form (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/14/NCT06263114/ICF_001.pdf